CLINICAL TRIAL: NCT05688267
Title: Effects of Continuous Mobility Training in Individuals With Prolonged Mechanical Ventilation : A Randomized Controlled Trial
Brief Title: Effects of Continuous Mobility Training in Prolonged Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Chi-Wen Lin, Physical Therapist, Taichung Tzu Chi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022CLin
Record Dates: First submitted 2022-12-29; First posted 2023-01-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Prolonged Mechanical Ventilation
Keywords: Mechanical Ventilator; Ventilator Weaning; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The continuous mobility training adopted grading exercise level, which was evaluated and implemented by physical therapists, and focused on continuous mobility training courses with different levels. At each stage, the participants were instructed to perform spontaneous breathing exercise, which were confirmed by the physical therapists. The five stages are half-lying on the bed, sitting at the bedside, sitting on the chair, standing and marching on spot.
  Interventions: Other: Continuous Mobility Training
- Control group (Placebo Comparator): Participants of control group formed the routine care group, received the routine mechanical ventilation weaning plan and underwent hand bicycle training. The physicians assessed the participants and appropriately adjusted the settings of the mechanical ventilation modules to gradually reduce the participants' dependence on mechanical ventilation. Hand bicycle training was conducted by nurse practitioners once a day. The participants' bedhead was raised, and the participants held the cycle ergometer with both hands once they could tolerate upright positions for 15-20 minutes. Training intensity was targeted at the level of symptom limitation, on the basis of a modified Borg scale rating of 3-5. Intermittent and short-term periods of rest were allowed for participants to achieve the goal of a total of 15-20 minutes exercise session.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Continuous Mobility Training — The continuous mobility training adopted 5 grading exercise level, which was evaluated and implemented by physical therapists, and focused on continuous mobility training courses with different levels. At each stage, the participants were instructed to perform spontaneous breathing exercise, which were confirmed by the physical therapists.
  Arms: Experimental group
Other: Usual Care — Participants of control group formed the routine care group, received the routine mechanical ventilation weaning plan and underwent hand bicycle training.
  Arms: Control group

SUMMARY:
Background: The exercise intervention can help participants with prolonged mechanical ventilation improve ventilator weaning; however, the content of exercise intervention is diverse and inconsistent.

Objective: This study aims to design the continuous mobility training and examine the clinical effects in participants with prolonged mechanical ventilation.

Methods: This prospective, single-center, concealed allocation, evaluator-blind, randomized control study divided participants transferred from the intensive care unit to the respiratory care center into two groups. The control group underwent the routine ventilator weaning plan and hand bicycle training, while the experimental group underwent routine ventilator weaning plan and continuous mobility training plan. The success rate of ventilator weaning, length of mechanical ventilation, length of stay at the respiratory care center, and total length of hospital stay were analyzed.

DETAILED DESCRIPTION:
The investigators designed a prospective, single-center, concealed allocation, evaluator-blind, intention-to-treat, randomized control study.

Participants This study was at the respiratory care center of a hospital in Taiwan. Individuals over 18 years of age, who used mechanical ventilation, were transferred from the intensive care unit to the respiratory care center for mechanical ventilation weaning, and were evaluated by a physician enrolled in the study. When a patient was eligible, the physician would conduct further examinations to ensure the suitability and safety of the participants, and the reasons for ineligibility for inclusion would be noted in the log.

Inclusion criteria:

1. Aged over 18 years, regardless of sex.
2. Use of mechanical ventilation and transfer from the intensive care unit to the respiratory care center for weaning.
3. Stable vital signs.
4. Ability to understand simple instructions and agree to participate in this research program after explanation.

Exclusion criteria:

1. Unconsciousness, severe cognitive impairment, or inability to follow instructions.
2. Severe heart failure (NYHA ≥ 3).
3. Diagnosis of terminal illness and undergoing palliative care.
4. Inability to receive exercise therapy due to physical conditions, fracture, lower limb surgery, acute thrombosis, open wounds, extracorporeal membrane oxygenation.
5. Assessment by other attending physician that the participant's condition, progression of disease course or treatment plan were not suitable for exercise therapy.

When the participants enrolled in the research, the trained research team members would explain the objectives and methods of the research to ensure that the participants' consent was fully informed. The participants had the right to withdraw from this research program at any time. If a participant was unwilling to participate or withdrew, they were excluded from this research program. A participant could only be enrolled after agreeing and signing the consent form. A randomized clinical trial design was adopted in this study. The participants were randomly divided into the experimental and control group in a one-to-one ratio. The research assistant placed the number plate in an opaque and sealed envelope to ensure concealed allocation. The order of allocation was randomized by the computer. The control group underwent the routine mechanical ventilation weaning plan and hand bicycle training, while the experimental group underwent the routine mechanical ventilation weaning plan and continuous mobility training. Owing to the nature of the exercise intervention, it is impossible to maintain blinding of the team members and participants. However, the physical therapists who evaluated the main outcome were separated from those who performed the therapy; thus, the evaluators were blinded. The content of the continuous mobility training program depended on the evaluation results and the physical responses of the participants. The treatment frequency of continuous mobility training was five times a week, once a day from Monday to Friday.

Intervention content Control group: Participants of control group formed the routine care group, received the routine mechanical ventilation weaning plan and underwent hand bicycle training. The physicians assessed the participants and appropriately adjusted the settings of the mechanical ventilation modules to gradually reduce the participants' dependence on mechanical ventilation. Hand bicycle training was conducted by nurse practitioners once a day. The participants' bedhead was raised, and the participants held the cycle ergometer with both hands once they could tolerate upright positions for 15-20 minutes. Training intensity was targeted at the level of symptom limitation, on the basis of a modified Borg scale rating of 3-5. Intermittent and short-term periods of rest were allowed for participants to achieve the goal of a total of 15-20 minutes exercise session.

Experimental group: Participants of the experimental group were given continuous mobility training in addition to the routine mechanical ventilation weaning plan. The protocol was divided into 5 levels - a modification from Dong et al. The physicians were responsible for evaluating whether the participants had any contraindications before and during enrolment. If any contraindication occurred at any time point, such as hypoxemia and other adverse events, the treatment would be terminated immediately. The continuous mobility training would be performed once a day from Monday to Friday. During the whole continuous mobility training process, the exercise progress would be increased gradually, depending on the tolerance and stability of the participants. The goal setting of each training exercise was that the participants could undergo the training for 20 minutes continuously.

The continuous mobility training adopted grading exercise level, which was evaluated and implemented by physical therapists, and focused on continuous mobility training courses with different levels. At each stage, the participants were instructed to perform spontaneous breathing exercise, which were confirmed by the physical therapists. In the first stage, the participants' bedhead were raised, and the trunk were kept upright on the bed. In sitting posture training, chest expansion training and deep breathing training was performed. The training goal was that the participants should be able to sit in bed for at least 20 minutes, and after training, the modified Borg scale rating of the participants should not exceed 7. If the participants could successfully complete the first stage of the exercise training, they would proceed to the next stage of exercise, and the training would be further upgraded to assisting the participants to sit at the bedside in an upright posture and perform sitting balance training. The physical therapists would provide minimal assistance or assistive devices according to the participants' conditions. The goal was to achieve tolerance for 20 minutes continuously with a modified RPE not exceeding 7 and no contraindications. In the third stage, the physical therapists would adopt appropriate strategies and assistive devices according to the participants' abilities and move the participants to chairs. The fourth stage was standing training. The participants could use assistive devices or other assistance to stand. The fifth stage was marching on spot. All exercise training was guided by the principle of maximum active participation of participants, with the goal of continuous completion of body movements and spontaneous breathing movements.

Termination conditions of continuous mobility training: The training would be terminated immediately if the participants had the following conditions:

1. Unstable vital signs: low blood oxygen concentration (SaO2 ≤ 90%) or shortness of breath (total respiratory rate > 35 beats/min).
2. Arrhythmia.
3. Severe dizziness.
4. Changes in consciousness.
5. Assessment by attending physician that the participant's condition, progression of disease course or treatment plan was not suitable for activities of exercise therapy.

After the intervention, the length of mechanical ventilation, length of stay in the respiratory care center, the success rate of mechanical ventilation weaning (weaning for more than 5 days), the total length of hospital stay and adverse events of two groups were recorded with evaluator-blind.

Data analysis All participants were included in the intention-to-treat analysis. The mean, standard deviation, and percentage of the participants' variables were used for descriptive statistics. Comparative analysis between the experimental group and the control group was performed according to all the effect variables. If the continuous variables conformed to normal distribution according to Shapiro-Wilk test, they were expressed as mean±standard deviation (mean±SD); otherwise, they were expressed as median (interquartile range). Categorical variables were expressed as percentage.

The evaluation records of the two groups of participants were compared, and continuous variables with normal distribution were compared by two sample independent t-test. When the data were not normally distributed, Mann-Whitney U test was used to compare the experimental group with the control group. Chi-square test was used to evaluate the differences in the categorical variables between the experimental group and the control group. To calculate the sample size for duration of mechanical ventilation, the investigators based the design on results found in Lai (2017) for a clinical trial. Considering a statistical power of 90% and alpha error of 0.5, the investigators found that the number of subjects should be 9 per group, totaling 18 participants. The statistical analysis software used was SPSS version 27.0, with 2-tailed p<.05 indicating statistical significance.

ELIGIBILITY:
Inclusion criteria:

1. Aged over 18 years, regardless of sex.
2. Use of mechanical ventilation and transfer from the intensive care unit to the respiratory care center for weaning.
3. Stable vital signs.
4. Ability to understand simple instructions and agree to participate in this research program after explanation.

Exclusion criteria:

1. Unconsciousness, severe cognitive impairment, or inability to follow instructions.
2. Severe heart failure (NYHA ≥ 3).
3. Diagnosis of terminal illness and undergoing palliative care.
4. Inability to receive exercise therapy due to physical conditions, fracture, lower limb surgery, acute thrombosis, open wounds, extracorporeal membrane oxygenation.
5. Assessment by other attending physician that the participant's condition, progression of disease course or treatment plan were not suitable for exercise therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
The success rate of ventilator weaning | up to 6 weeks
  The success rate of ventilator weaning

SECONDARY OUTCOMES:
The length of mechanical ventilation | up to 6 weeks
  The length of mechanical ventilation
The length of stay at the respiratory care center | up to 6 weeks
  The length of stay at the respiratory care center
The total length of hospital stay | up to 12 weeks
  The total length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Wen Lin, Study Chair — Taichung Tzu Chi Hospital
Locations (1):
- Taichung Tzu Chi Hospital, Taichang, Taiwan

IPD SHARING:
Plan to Share IPD: No
Weaning from Prolonged Mechanical Ventilation

REFERENCES:
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Powers SK, Wiggs MP, Sollanek KJ, Smuder AJ. Ventilator-induced diaphragm dysfunction: cause and effect. Am J Physiol Regul Integr Comp Physiol. 2013 Sep;305(5):R464-77. doi: 10.1152/ajpregu.00231.2013. Epub 2013 Jul 10. PMID 23842681
- [Background] Thomas P, Baldwin C, Bissett B, Boden I, Gosselink R, Granger CL, Hodgson C, Jones AY, Kho ME, Moses R, Ntoumenopoulos G, Parry SM, Patman S, van der Lee L. Physiotherapy management for COVID-19 in the acute hospital setting: clinical practice recommendations. J Physiother. 2020 Apr;66(2):73-82. doi: 10.1016/j.jphys.2020.03.011. Epub 2020 Mar 30. PMID 32312646
- [Background] Ntoumenopoulos G. Rehabilitation during mechanical ventilation: Review of the recent literature. Intensive Crit Care Nurs. 2015 Jun;31(3):125-32. doi: 10.1016/j.iccn.2015.02.001. Epub 2015 May 27. PMID 26026495
- [Background] Rose L, McGinlay M, Amin R, Burns KE, Connolly B, Hart N, Jouvet P, Katz S, Leasa D, Mawdsley C, McAuley DF, Schultz MJ, Blackwood B. Variation in Definition of Prolonged Mechanical Ventilation. Respir Care. 2017 Oct;62(10):1324-1332. doi: 10.4187/respcare.05485. Epub 2017 Jun 13. PMID 28611229
- [Background] Rojek-Jarmula A, Hombach R, Krzych LJ. APACHE II score cannot predict successful weaning from prolonged mechanical ventilation. Chron Respir Dis. 2017 Aug;14(3):270-275. doi: 10.1177/1479972316687100. Epub 2017 Feb 24. PMID 28774204
- [Background] Damuth E, Mitchell JA, Bartock JL, Roberts BW, Trzeciak S. Long-term survival of critically ill patients treated with prolonged mechanical ventilation: a systematic review and meta-analysis. Lancet Respir Med. 2015 Jul;3(7):544-53. doi: 10.1016/S2213-2600(15)00150-2. Epub 2015 May 20. PMID 26003390
- [Background] Cox CE, Carson SS, Holmes GM, Howard A, Carey TS. Increase in tracheostomy for prolonged mechanical ventilation in North Carolina, 1993-2002. Crit Care Med. 2004 Nov;32(11):2219-26. doi: 10.1097/01.ccm.0000145232.46143.40. PMID 15640633
- [Background] Schreiber A, Bertoni M, Goligher EC. Avoiding Respiratory and Peripheral Muscle Injury During Mechanical Ventilation: Diaphragm-Protective Ventilation and Early Mobilization. Crit Care Clin. 2018 Jul;34(3):357-381. doi: 10.1016/j.ccc.2018.03.005. PMID 29907270
- [Background] Mendez-Tellez PA, Needham DM. Early physical rehabilitation in the ICU and ventilator liberation. Respir Care. 2012 Oct;57(10):1663-9. doi: 10.4187/respcare.01931. PMID 23013903
- [Background] Kim WY, Lim CM. Ventilator-Induced Diaphragmatic Dysfunction: Diagnosis and Role of Pharmacological Agents. Respir Care. 2017 Nov;62(11):1485-1491. doi: 10.4187/respcare.05622. Epub 2017 Jul 11. PMID 28698263
- [Background] Penuelas O, Frutos-Vivar F, Fernandez C, Anzueto A, Epstein SK, Apezteguia C, Gonzalez M, Nin N, Raymondos K, Tomicic V, Desmery P, Arabi Y, Pelosi P, Kuiper M, Jibaja M, Matamis D, Ferguson ND, Esteban A; Ventila Group. Characteristics and outcomes of ventilated patients according to time to liberation from mechanical ventilation. Am J Respir Crit Care Med. 2011 Aug 15;184(4):430-7. doi: 10.1164/rccm.201011-1887OC. PMID 21616997
- [Background] Sansone GR, Frengley JD, Vecchione JJ, Manogaram MG, Kaner RJ. Relationship of the Duration of Ventilator Support to Successful Weaning and Other Clinical Outcomes in 437 Prolonged Mechanical Ventilation Patients. J Intensive Care Med. 2017 May;32(4):283-291. doi: 10.1177/0885066615626897. Epub 2016 Jan 20. PMID 26792815
- [Background] Ding N, Zhang Z, Zhang C, Yao L, Yang L, Jiang B, Wu Y, Jiang L, Tian J. What is the optimum time for initiation of early mobilization in mechanically ventilated patients? A network meta-analysis. PLoS One. 2019 Oct 7;14(10):e0223151. doi: 10.1371/journal.pone.0223151. eCollection 2019. PMID 31589642
- [Background] McWilliams D, Jones C, Atkins G, Hodson J, Whitehouse T, Veenith T, Reeves E, Cooper L, Snelson C. Earlier and enhanced rehabilitation of mechanically ventilated patients in critical care: A feasibility randomised controlled trial. J Crit Care. 2018 Apr;44:407-412. doi: 10.1016/j.jcrc.2018.01.001. Epub 2018 Jan 4. PMID 29331668
- [Background] Morris PE, Berry MJ, Files DC, Thompson JC, Hauser J, Flores L, Dhar S, Chmelo E, Lovato J, Case LD, Bakhru RN, Sarwal A, Parry SM, Campbell P, Mote A, Winkelman C, Hite RD, Nicklas B, Chatterjee A, Young MP. Standardized Rehabilitation and Hospital Length of Stay Among Patients With Acute Respiratory Failure: A Randomized Clinical Trial. JAMA. 2016 Jun 28;315(24):2694-702. doi: 10.1001/jama.2016.7201. PMID 27367766
- [Background] Camargo Pires-Neto R, Fogaca Kawaguchi YM, Sayuri Hirota A, Fu C, Tanaka C, Caruso P, Park M, Ribeiro Carvalho CR. Very early passive cycling exercise in mechanically ventilated critically ill patients: physiological and safety aspects--a case series. PLoS One. 2013 Sep 9;8(9):e74182. doi: 10.1371/journal.pone.0074182. eCollection 2013. PMID 24040200
- [Background] Chang MY, Chang LY, Huang YC, Lin KM, Cheng CH. Chair-sitting exercise intervention does not improve respiratory muscle function in mechanically ventilated intensive care unit patients. Respir Care. 2011 Oct;56(10):1533-8. doi: 10.4187/respcare.00938. Epub 2011 Apr 19. PMID 21513602
- [Background] Dong Z, Yu B, Zhang Q, Pei H, Xing J, Fang W, Sun Y, Song Z. Early Rehabilitation Therapy Is Beneficial for Patients With Prolonged Mechanical Ventilation After Coronary Artery Bypass Surgery. Int Heart J. 2016;57(2):241-6. doi: 10.1536/ihj.15-316. Epub 2016 Mar 11. PMID 26973269
- [Background] Lai CC, Chou W, Chan KS, Cheng KC, Yuan KS, Chao CM, Chen CM. Early Mobilization Reduces Duration of Mechanical Ventilation and Intensive Care Unit Stay in Patients With Acute Respiratory Failure. Arch Phys Med Rehabil. 2017 May;98(5):931-939. doi: 10.1016/j.apmr.2016.11.007. Epub 2016 Dec 13. PMID 27979608
- [Background] Verceles AC, Wells CL, Sorkin JD, Terrin ML, Beans J, Jenkins T, Goldberg AP. A multimodal rehabilitation program for patients with ICU acquired weakness improves ventilator weaning and discharge home. J Crit Care. 2018 Oct;47:204-210. doi: 10.1016/j.jcrc.2018.07.006. Epub 2018 Jul 11. PMID 30025227
- [Background] Sollanek KJ, Smuder AJ, Wiggs MP, Morton AB, Koch LG, Britton SL, Powers SK. Role of intrinsic aerobic capacity and ventilator-induced diaphragm dysfunction. J Appl Physiol (1985). 2015 Apr 1;118(7):849-57. doi: 10.1152/japplphysiol.00797.2014. Epub 2015 Jan 8. PMID 25571991
- [Background] Yang PH, Wang CS, Wang YC, Yang CJ, Hung JY, Hwang JJ, Wang TH, Chuang IC, Huang MS. Outcome of physical therapy intervention on ventilator weaning and functional status. Kaohsiung J Med Sci. 2010 Jul;26(7):366-72. doi: 10.1016/S1607-551X(10)70060-7. PMID 20638039
- [Background] Clarissa C, Salisbury L, Rodgers S, Kean S. Early mobilisation in mechanically ventilated patients: a systematic integrative review of definitions and activities. J Intensive Care. 2019 Jan 17;7:3. doi: 10.1186/s40560-018-0355-z. eCollection 2019. PMID 30680218
- [Background] Costa DK, White MR, Ginier E, Manojlovich M, Govindan S, Iwashyna TJ, Sales AE. Identifying Barriers to Delivering the Awakening and Breathing Coordination, Delirium, and Early Exercise/Mobility Bundle to Minimize Adverse Outcomes for Mechanically Ventilated Patients: A Systematic Review. Chest. 2017 Aug;152(2):304-311. doi: 10.1016/j.chest.2017.03.054. Epub 2017 Apr 21. PMID 28438605
- [Background] TEAM Study Investigators; Hodgson C, Bellomo R, Berney S, Bailey M, Buhr H, Denehy L, Harrold M, Higgins A, Presneill J, Saxena M, Skinner E, Young P, Webb S. Early mobilization and recovery in mechanically ventilated patients in the ICU: a bi-national, multi-centre, prospective cohort study. Crit Care. 2015 Feb 26;19(1):81. doi: 10.1186/s13054-015-0765-4. PMID 25715872
- [Background] Patman SM, Dennis DM, Hill K. Exploring the capacity to ambulate after a period of prolonged mechanical ventilation. J Crit Care. 2012 Dec;27(6):542-8. doi: 10.1016/j.jcrc.2011.12.020. Epub 2012 Mar 14. PMID 22421005
- [Background] Hill K, Dennis DM, Patman SM. Relationships between mortality, morbidity, and physical function in adults who survived a period of prolonged mechanical ventilation. J Crit Care. 2013 Aug;28(4):427-32. doi: 10.1016/j.jcrc.2013.02.012. Epub 2013 Apr 22. PMID 23618778
- [Background] Goddard SL, Lorencatto F, Koo E, Rose L, Fan E, Kho ME, Needham DM, Rubenfeld GD, Francis JJ, Cuthbertson BH. Barriers and facilitators to early rehabilitation in mechanically ventilated patients-a theory-driven interview study. J Intensive Care. 2018 Jan 23;6:4. doi: 10.1186/s40560-018-0273-0. eCollection 2018. PMID 29403646
- [Background] Nydahl P, Ruhl AP, Bartoszek G, Dubb R, Filipovic S, Flohr HJ, Kaltwasser A, Mende H, Rothaug O, Schuchhardt D, Schwabbauer N, Needham DM. Early mobilization of mechanically ventilated patients: a 1-day point-prevalence study in Germany. Crit Care Med. 2014 May;42(5):1178-86. doi: 10.1097/CCM.0000000000000149. PMID 24351373
- [Background] Chiang LL, Wang LY, Wu CP, Wu HD, Wu YT. Effects of physical training on functional status in patients with prolonged mechanical ventilation. Phys Ther. 2006 Sep;86(9):1271-81. doi: 10.2522/ptj.20050036. PMID 16959675
- [Background] Chen S, Su CL, Wu YT, Wang LY, Wu CP, Wu HD, Chiang LL. Physical training is beneficial to functional status and survival in patients with prolonged mechanical ventilation. J Formos Med Assoc. 2011 Sep;110(9):572-9. doi: 10.1016/j.jfma.2011.07.008. Epub 2011 Sep 8. PMID 21930067
- [Background] Elkins M, Dentice R. Inspiratory muscle training facilitates weaning from mechanical ventilation among patients in the intensive care unit: a systematic review. J Physiother. 2015 Jul;61(3):125-34. doi: 10.1016/j.jphys.2015.05.016. Epub 2015 Jun 16. PMID 26092389
- [Background] Clini EM, Crisafulli E, Antoni FD, Beneventi C, Trianni L, Costi S, Fabbri LM, Nava S. Functional recovery following physical training in tracheotomized and chronically ventilated patients. Respir Care. 2011 Mar;56(3):306-13. doi: 10.4187/respcare.00956. Epub 2010 Nov 16. PMID 21235844
- [Background] Martin UJ, Hincapie L, Nimchuk M, Gaughan J, Criner GJ. Impact of whole-body rehabilitation in patients receiving chronic mechanical ventilation. Crit Care Med. 2005 Oct;33(10):2259-65. doi: 10.1097/01.ccm.0000181730.02238.9b. PMID 16215380